CLINICAL TRIAL: NCT01172470
Title: Phase II Trial of Pemetrexed-Based Induction Chemotherapy Followed by Concomitant Chemoradiotherapy in Previously Irradiated Head and Neck Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13881B
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer
Keywords: Recurrent head and neck cancer; larynx, lip, oral cavity and pharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases; Lymphoid Interstitial Pneumonia | interventions — Gemcitabine; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gemcitabine — 4 doses of induction chemotherapy every 2weeks, IV (in the vein)
Drug: Pemetrexed — Induction Chemotherapy:
  4 doses of induction chemotherapy every 2weeks(Days 1, 15, 28, and 42), through an infusion for approximately 10 minutes.
  Chemoradiotherapy:
  Day 1,22, and 43through IV infusion over a period of 10 minutes
Drug: Carboplatin — Chemoradiotherapy:
  Day 1, 22 and 4 through IV infusion over a period of 1 hour.

SUMMARY:
The purpose of this study is to determine 1-year survival of previously irradiated Head and Neck cancer (HNC) patients with loco-regional recurrent disease treated with induction chemotherapy with pemetrexed and gemcitabine followed concomitant pemetrexed, carboplatin and daily radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All previously irradiated patients with recurrent head and neck cancer with no clinically measurable distant disease or those patients in whom distant disease was of low volume and local and regional palliation is clinically warranted. Low volume metastatic disease is defined as asymptomatic or minimally symptomatic disease that, according to physician judgment and without therapy for locoregionally recurrent disease, is unlikely to effect the subject's quality or quantity of life.
* Histologic or cytological documentation of recurrent head and neck cancer requiring regional therapy.
* Prior radiation therapy completed > 4 months before to study entry, if patients have recovered from all side effects grade 1.
* Predominance of disease that is amenable to radiotherapy.
* Measurable disease prior to induction chemotherapy.
* Age >18 years
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky > 70%).
* Patients must have normal organ and marrow function as defined below:

Leukocytes >3,000/ul Absolute neutrophil count >1,500/ul Platelets >100,000/ul Total bilirubin < 1.5X institutional upper limit of normal AST (SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal Creatinine Clearance (CrCl) > 45 mL/min

The standard Cockcroft and Gault formula (based on actual weight) or the measured glomerular filtration rate (GFR) using the appropriate radiolabeled method (51-CrEDTA or Tc99m-DTPA) must be used to calculate CrCl for enrollment or dosing. The same method used at baseline should be used throughout the study. Insufficient numbers of patients have been studied with creatinine clearance <45 mL/min to give a dose recommendation. Therefore, pemetrexed should not be administered to patients whose creatinine clearance is <45 mL/min.

Although ibuprofen and other non-steroidal inflammatory drugs (NSAID) can be administered with pemetrexed in patients with normal renal function (creatinine clearance 80 mL/min), caution should be used when administering NSAID concurrently with pemetrexed to patients with mild to moderate renal insufficiency (creatinine clearance from 45 to 79 mL/min). Patients with mild to moderate renal insufficiency should avoid taking NSAID with short elimination half lives (e.g. ibuprofen) for a period of 2 days before, the day of, and 2 days following administration of pemetrexed. In the absence of data regarding potential interaction between pemetrexed and NSAID with longer half lives, all patients taking these NSAID should interrupt dosing for at least 5 days before, the day of, and 2 days following pemetrexed administration. If concomitant administration of an NSAID is necessary, patients should be monitored closely for toxicity, especially myelosuppression, renal, and gastrointestinal toxicity.

* The presence of a significant infection or another severe complicating medical illness may constitute a contraindication to entrance on this protocol.
* Pregnancy is an absolute contraindication for this treatment protocol.
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow vitamins and dexamethasone or willingness to use a feeding tube to ingest these agents

Exclusion Criteria:

Previously untreated patients are not eligible

Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.

Patients may not be receiving any other investigational agents.

History of allergic reactions attributed to compounds of similar chemical composition agents used in the study.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Primary objective is to determine 1-year survival of previously irradiated Head/Neck Cancer patients with loco-regional recurrent disease treated with induction chemotherapy with pemetrexed and gemcitabine followed by concomitant pemetrexed, carboplat | 1-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Principal Investigator — The University of Chicago Medical Center
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Ziliak D, O'Donnell PH, Im HK, Gamazon ER, Chen P, Delaney S, Shukla S, Das S, Cox NJ, Vokes EE, Cohen EE, Dolan ME, Huang RS. Germline polymorphisms discovered via a cell-based, genome-wide approach predict platinum response in head and neck cancers. Transl Res. 2011 May;157(5):265-72. doi: 10.1016/j.trsl.2011.01.005. Epub 2011 Feb 8. PMID 21497773
- See also: (The University of Chicago Comprehensive Cancer Center Web page. — http://uccrc.uchicago.edu/